CLINICAL TRIAL: NCT02073474
Title: An Observational Post-Marketing Safety Registry Of Patients Who Have Been Prescribed Sativex®
Brief Title: An Observational Post-Marketing Safety Registry of Sativex®
Status: Completed | Type: Observational
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: GWSR10128
Record Dates: First submitted 2014-02-21; First posted 2014-02-27 (Estimated); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Multiple Sclerosis; Diabetes; Cancer; Neuropathic Pain
Keywords: cannabinoids; Sativex; THC; delta-9-tetrahydrocannabinol; cannabidiol; CBD; Registry; Safety; MS
MeSH Terms: conditions — Multiple Sclerosis; Diabetes Mellitus; Neoplasms; Neuralgia; Marijuana Abuse | interventions — nabiximols

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Sativex® users: UK: All patients and who are prescribed Sativex®. Germany and Sweden: Patients who are prescribed Sativex® from selected specialist neurology centres.
  Interventions: Drug: Sativex®

INTERVENTIONS:
Drug: Sativex® — Contains delta-9-tetrahydrocannabinol (THC), 27 mg/mL; cannabidiol (CBD), 25 mg/mL; in ethanol:propylene glycol (50:50) excipients, with peppermint oil (0.05%) flavouring. Each actuation delivers THC 2.7 mg and CBD 2.5 mg.
  Other Names: Nabiximols; GWP42001; THC/CBD spray

SUMMARY:
The purpose of this registry is to monitor safety outcomes of patients who are receiving Sativex® for Multiple Sclerosis (MS) spasticity and for off-label indications in the United Kingdom (UK), Germany and Sweden.

DETAILED DESCRIPTION:
The objectives of this multi-centre, observational program are to evaluate the long-term safety of Sativex® with special regard to the following:

* The potential for addiction, abuse and misuse for illegal purposes
* The potential for long-term psychiatric effects including suicidality and psychosis
* The potential for mood changes / psychological effects (such as confusion / disorientation)
* The potential for memory impairment
* The effect on driving ability
* The potential for falls
* The use of MS concomitant medications

All physicians who are prescribing Sativex® in the UK and those from specialist neurology centres in Germany and Sweden will be invited to participate in the registry and will be provided with information regarding the background and objectives of the study. The prescribing physician will be asked to enter the following information via electronic Case Report Forms (CRF) at 6 monthly intervals for up to 24 months for any one patient:

Sativex® Use:

* Was Sativex® prescribed for Spasticity in MS? (Yes/No). If no, specify then indication for prescribing Sativex®
* Year of Spasticity diagnosis (Germany/Sweden only)
* Sativex® start date
* Sativex® daily dose (average, minimum and maximum)
* Date of last prescription
* Is Sativex® providing worthwhile benefit? (Yes/ No/ Don't Know)
* Has Sativex® been stopped permanently? (Yes /No). If yes, reason for stopping is to be provided.
* Sativex® stop date

Adverse Events (AE):

* Have any clinically significant adverse events been reported for this patient since they started taking Sativex® (initial record); did any clinically significant adverse events occur, or were ongoing, during this period (follow-up records) (If yes, the details are recorded on an AE form)
* Has the patient sought medical attention because of a fall related injury; since they started taking Sativex® (initial record); during this period (follow-up records) (If yes, the details are recorded on an AE form)
* Has the patient experienced any suicidal thoughts or attempted suicide; since they started taking Sativex® (initial record); during this period (follow-up records) (If yes, the details are recorded on an AE form)
* Has the patient experienced any other significant psychiatric or psychotic events; since they started taking Sativex® (initial record); during this period (follow-up records) (If yes, the details are recorded on an AE form)
* Has the patient reported any change in their driving ability; since they started taking Sativex® (initial record); during this period (follow-up records)

  * Improved
  * No change
  * Deteriorated
  * Not appropriate

Supporting Information:

* Medical History relevant to adverse events
* What other Spasticity medications have previously been used and are now stopped permanently (baclofen, tizanidine, benzodiazepines, gabapentin, botulinum toxin) (Germany/Sweden only)
* Changes to other MS symptom medications; since they started taking Sativex® (initial record); during this period (follow-up records)?

Survival status:

* Is the patient currently alive? If no, date of death and cause of death.
* Was the death due to suicide (Yes/No)

Paper CRF will also be available and will subsequently be entered into the electronic CRF database.

The data from the Registry will be analysed descriptively and collated into summary tables and listings.

A Registry report based upon the data summaries will be included within the Periodic Safety Update Reports for Sativex® and the results will be submitted to the appropriate Regulatory Agencies within 60 days of the data summaries tables and listings becoming available.

Each six monthly report and the data tables and listings will be reviewed by an independent Sativex® Registry Advisory Board and a summary overview will be prepared by the committee.

A final Registry report will be assembled within 180 days of the final study data being available.

Any significant safety issues identified will be communicated to the relevant Regulatory Agencies immediately.

ELIGIBILITY:
Inclusion Criteria:

* All patients who are prescribed Sativex® in the UK
* Patients who are prescribed Sativex® from selected specialist neurology centres in Germany and Sweden.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who are prescribed Sativex® in the UK and patients who are prescribed Sativex® from selected specialist neurology centres in Germany and Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 978 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Incidence rates of adverse events. | Participants will be followed for the duration of Sativex treatment, an expected average of 2 years.
  The number of treatment-emergent adverse events was recorded. The incidence rate (number of patients divided by the total patient-years exposure to Sativex®) for each adverse event is presented.

SECONDARY OUTCOMES:
Average daily number of sprays of Sativex® used. | Participants will be followed for the duration of Sativex treatment, an expected average of 2 years.
  The average daily dose of Sativex® was recorded and is presented.
Number of patients experiencing fall-related injuries requiring medical attention. | Participants will be followed for the duration of Sativex treatment, an expected average of 2 years.
  Patients were asked if they had sought medical attention because of a fall-related injury; since they started taking Sativex® (initial record); during this period (follow-up records). The number of patients answering 'yes' is presented.
Number of patients experiencing a change in driving ability. | Participants will be followed for the duration of Sativex treatment, an expected average of 2 years.
  Patients were asked to report any change in their driving ability; since they started taking Sativex® (initial record); during this period (follow-up records). The markers were: Improved, No change, Deteriorated, Not appropriate. The number of patients for each marker is presented.
Number of patients experiencing suicidal thoughts or attempts. | Participants will be followed for the duration of Sativex treatment, an expected average of 2 years.
  Patients were asked if they had experienced any suicidal thoughts or attempted suicide; since they started taking Sativex® (initial record); during this period (follow-up records). The number of patients answering 'yes' is presented.
Number of patients experiencing significant psychiatric or psychotic events other than suicidality. | Participants will be followed for the duration of Sativex treatment, an expected average of 2 years.
  Patients were asked if they had experienced any significant psychiatric or psychotic events other than suicidality; since they started taking Sativex® (initial record); during this period (follow-up records). The number of patients answering 'yes' is presented.
Incidence of patient deaths. | Participants will be followed for the duration of Sativex treatment, an expected average of 2 years.
  The incidence of treatment-emergent deaths was recorded and the number of patient deaths is presented.
Number of patients receiving worthwhile benefit from Sativex®. | Participants will be followed for the duration of Sativex treatment, an expected average of 2 years.
  Patients were asked if Sativex® was providing worthwhile benefit. The number of patients answering 'yes' at one or more time points is presented.
Number of MS patients discontinuing anti-spasticity medications. | Participants will be followed for the duration of Sativex treatment, an expected average of 2 years.
  MS patients were asked what other anti-spasticity medications that have previously been used are now stopped permanently; since they started taking Sativex® (initial record); during this period (follow-up records). The number of patients for each discontinued medication is presented.
Number of MS patients discontinuing medications for MS symptoms other than anti-spasticity medications. | Participants will be followed for the duration of Sativex treatment, an expected average of 2 years.
  MS patients were asked what medications for MS symptom other than anti-spasticity medications that have previously been used are now stopped permanently; since they started taking Sativex® (initial record); during this period (follow-up records). The number of patients for each discontinued medication is presented.